CLINICAL TRIAL: NCT07064239
Title: Effect of Cooling Vest on Fatigue and Spatiotemporal Gait Parameters in Multiple Sclerosis Patients
Brief Title: Effect of Cooling Vest in Multiple Sclerosis Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Khalil essa ibrahim, Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.Rec/012/005788
Record Dates: First submitted 2025-06-20; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A placebo group (Placebo Comparator): include A 15 individuals with relapsing-remitting MS performed 30 minutes of aerobic exercise (upper- and lower-extremity ergometry and treadmill ambulation) without wearing cooling vest, followed by unstructured physical activity. 15 participants completed the intervention and posttest follow-up. quality of life (measured with the Multiple Sclerosis Quality of Life-54; MSQOL-54) were assessed. Participants completed 27.9 minutes of exercise per session, session will done for three sessions of aerobic exercise and Frenkel Coordination Exercises per week for 6 weeks.
  Interventions: Other: Aerobic exercises
- Group B cooling vest group (Experimental): include A 15 individuals with relapsing-remitting MS performed 30 minutes of aerobic exercise (upper- and lower-extremity ergometry and treadmill ambulation) with wearing cooling vest, followed by unstructured physical activity. Eight participants completed the intervention and posttest follow-up. quality of life (measured with the Multiple Sclerosis Quality of Life-54; MSQOL-54) were assessed. Participants completed 27.9 minutes of exercise per session, session will done for three sessions of aerobic exercise and Frenkel Coordination Exercises per week for 6 weeks.
  Interventions: Device: cooling vest; Other: Aerobic exercises

INTERVENTIONS:
Device: cooling vest — Cooling vest :
  It is one of cooling methods proposed to improve exercise performance in MS by reducing one's core and/or skin temperature before taking on physical work
  Arms: Group B cooling vest group
Other: Aerobic exercises — aerobic exercise as any activity that uses large muscle groups, can be maintained continuously and is rhythmic in nature. As the name implies, muscle groups activated by this type of exercise rely on aerobic metabolism to extract energy in the form of adenosine triphosphate (ATP) from amino acids, carbohydrates and fatty acids. Examples of aerobic exercise include cycling, dancing, hiking, jogging/long distance running, swimming and walking

SUMMARY:
This study is prospective, randomized controlled trail that will be conducted to investigate the effect of cooling therapy on fatigue and gait in patient with multiple sclerosis(MS).

DETAILED DESCRIPTION:
Thirty patients from both sexes will be enrolled in this study. They will be assigned into two equal groups (study and control groups). Patients will be diagnosed as MS patients based on careful clinical evaluation by the neurologist and magnetic resonance imaging (MRI) of the brain. The patients will be recruited from the faculty of Physical Therapy, Cairo University, and El Kasr El Ainy hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Thirty MS patients of both sexes.
* Age of patients ranges from 20 to 40 years.
* NOT less than 8 months since Symptoms onset.
* The body mass index ranged (BMI) from 20 - 24.5 Kg/m2 .
* The grade of The muscle tone of the affected limbs muscles ranged from 1
* to 2 grade according to Modified Ashower scale of muscle tone
* All the patients are medically stable.
* Patients have intact sensations (deep & superficial).

Exclusion Criteria:

* Other neurological and orthopedic impairments in upper or lower limb.
* Having visual and hearing problems.
* Inability to sit independently on a chair.
* Impaired cognition and impaired comprehension and ideomotor apraxia.
* History of endogenous depression or severe psychiatric disorders.
* Severe neglect, and major medical problems or comorbidities that will influence upper or lower extremity usage or cause severe pain.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2025-07-08 (Estimated)

PRIMARY OUTCOMES:
fatigue | At baseline and re assessed 6 weeks later.
  assessed by Fatigue Severity Scale(FSS): FSS is designed to measure fatigue in a single dimension using the nine items, which represent a single scale. Each FSS item consists of statements that are scored on a seven-point Likert type scale ranging from 1 ("strongly disagree") to 7 ("strongly agree"). The mean of the nine item scores is used as the FSS score, which ranges from 1 to 7. However, some studies have calculated an FSS score as the sum of all nine items, ranging from 9 to 63.The unit of measurement is points.
gait parameter (Gait Speed) | At baseline and re assessed 6 weeks later.
  kinovea software used for assessment:
  • The unit of measurement for gait speed is meter/second (m/sec)
gait parameters: Stride Length and Stride Length | At baseline and re assessed 6 weeks later.
  kinovea software used for assessment:
  • The unit of measurement for Stride Length and Stride Length is centimeter (cm)
gait parameter (Double Support) | At baseline and re assessed 6 weeks later.
  kinovea software used for assessment:
  • The unit of measurement for Double Support is seconds (sec)

SECONDARY OUTCOMES:
functional capacity | At baseline and re assessed 6 weeks later.
  functional capacity assessed using six minute walk test(meters/minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt